CLINICAL TRIAL: NCT05046067
Title: Feasibility Study of Anatomical Modeling for Image Guided Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-1189; NCI-2021-06616 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1189 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-07-18; First posted 2021-09-16 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-07

CONDITIONS: Lung Neoplasm
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (CT) (Experimental): Patients undergo 4 CT scans during standard of care surgery.
  Interventions: Procedure: Computed Tomography; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Therapeutic Conventional Surgery — Undergo surgery per standard of care

SUMMARY:
This clinical trial assesses the feasibility of creating a 3 dimensional (D) model of the lung and lung nodule(s) from computed tomography (CT) scan images performed during lung surgery. Unlike solid organs (like the kidney, brain, and liver), the lung changes shape (they inflate when a person breathe in and collapse when they breathe out). This makes it difficult to predict where, exactly, the tumor(s) will be on the lungs during surgery. A 3D model may help surgeons better predict where the location of the tumor(s) will be during surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the feasibility of developing an anatomical model to predict the location of the tumor in a deflated lung to assist in guidance during lung surgery.

SECONDARY OBJECTIVES:

I. Develop a registration technique to register the tumor onto the 2D/3D optical image obtained during surgery.

II. Determine the accuracy of mapping major segmental vasculature and bronchial structures onto 2D/3D optical images obtained during surgery.

OUTLINE:

Patients undergo 4 CT scans during standard of care surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have previous CT images demonstrating a lung mass or masses amenable to lung resection (open or minimally invasive)
* Patient is scheduled for surgical resection in a room equipped with intraoperative CT
* Patient must sign informed consent, with risks and benefits of CT imaging explained
* Patients with lung tumors >= 1cm to =< 3 cm based on preoperative CT scan. (Patients with lung tumors from < 1 cm or > 3 cm will be reviewed and approved for inclusion on an individual assessment by clinical collaborators)

Exclusion Criteria:

* Pediatric patients less than 18 years of age
* Patients who have undergone previous ipsilateral thoracic surgery, sclerotherapy, or radiation therapy as intraoperative adhesions may limit lung collapse intraoperatively
* Patients who received neoadjuvant immunotherapy
* Women who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Feasibility of anatomical modeling for image guided thoracic surgery | Up to 1 year
  The geometrical accuracy of the models for localizing the tumor will be quantified. The study is feasible if tumors for all 10 patients can be located with accuracy of within 1 cm or less. Anatomical modeling for image guided thoracic surgery will be considered feasible if researchers are able to determine the location of the tumor in a deflated lung to within the accuracy required by the surgeon for clinical use.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Rajaram, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/67/NCT05046067/ICF_000.pdf